CLINICAL TRIAL: NCT01317836
Title: PET-CT in Diagnosis of Pancreatic Cystic Neoplasms
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: PANCYST
Record Dates: First submitted 2011-03-16; First posted 2011-03-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Neoplasms; Pancreatic Cancer
Keywords: pancreatic cystic lesion; PET; PET-CT; diagnosis
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients having pancreatic cystic lesion

SUMMARY:
Preoperative diagnosis of pancreatic cystic lesions remains a difficult problem in clinical practice. At present, the treatment planning in pancreatic cystic neoplasms is significantly restricted by the limited preoperative diagnosis. Ultrasonography (US), multidetector computed tomography (MDCT) and magnetic resonance imaging (MRI) are the conventional modalities in imaging of pancreatic cystic neoplasms, but by these methods the diagnostic accuracy still remains compromised. Furthermore, recently encouraging results have been obtained in pancreatic cystic neoplasms using 18F-fluoro-2-deoxyglucose positron emission tomography (18F-FDG-PET) The aim of the current project is to evaluate the possibility to enhance the diagnostic accuracy by using the combined 18F-FDG-PET-CT imaging in patients with pancreatic cystic neoplasms by combining PET-CT with MRI and MDCT.

DETAILED DESCRIPTION:
Today, in clinical practice the diagnosis pancreatic cystic neoplasms are based on MDCT, MRI and ERCP followed by surgical exploration. The information gained by conventional imaging modalities is restricted to the morphological details, which usually is insufficient for the definitive staging of the pancreatic cystic neoplasms. Based on these previous studies, it seems that PET especially combined with CT modality could improve the diagnostic accuracy of the pancreatic cystic lesions.

So far, there are only few cases published concerning the role of 18F-FDG-PET-CT in the differential diagnosis of cystic pancreatic lesions. Therefore, more studies are needed to determine the role of combined 18F-FDG-PET-CT in the diagnosis of pancreatic cystic lesions.

The aim of the current project is to evaluate the possibility to enhance the diagnostic accuracy by using the combined 18F-FDG-PET-CT imaging in patients with pancreatic cystic neoplasms by combining PET-CT with MRI and MDCT.

The study consists of 20-30 patients with pancreatic cystic neoplasms. The patients enrolled in the study will be imaged by MDCT, MRI combined with magnetic resonance cholangiopancreatography (MRCP), endoscopic retrograde cholangiopancreatography (ERCP) and 18F-FDG-PET-CT followed by surgery or follow-up. The data will be collected between 2011 and 2013.

ELIGIBILITY:
Inclusion Criteria:

* suspicion of pancreatic cystic neoplasm using US, MDCT, MRI and/or ERCP
* laparotomy planned because of the lesion
* signed informed consent

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study subjects will be recruited from gastroenterological surgery department of Turku University Hospital with clinical suspicion of pancreatic cystic neoplasm.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Predictive Value of PET/CT imaging for Identifying Malignant and Benign Pancreatic Cystic Lesions | 1 mo
  To determine sensitivities, specificities, accuracy and positive/negative predictive values of PET/CT imaging for differentiating malignant and benign cystic lesions in patients who are to undergo surgical resection.

SECONDARY OUTCOMES:
To compare PET/CT to ERCP, MDCT and MRI-MRCP | 1 mo

CONTACTS AND LOCATIONS:
Overall Officials: Saila Kauhanen, PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku University Hospital, Turku, Finland